CLINICAL TRIAL: NCT02836145
Title: Biomolecular Messages Associated With the Differentiation of Human Induced Pluripotent Stem Cells to Skeletal Muscle Progenitor Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: NTU-REC-201603059RINA
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Female Urinary Incontinence and Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: Differentiation of hiPSCs to skeletal muscle progenitors

SUMMARY:
Female urinary incontinence and pelvic organ prolapse are common diseases especially in aged women that frequently cause urogenital infection, voiding difficulty, urinary retention, pelvic pain, constipation, and coital difficulty, as well as impact the quality of life of women. Risk factors of the above diseases include pregnancy, vaginal delivery, and menopausal status. Despite playing a crucial role in the pathophysiology of the above diseases, the urogenital skeletal muscular dysfunction cannot be fully corrected via the current treatment modalities.

The human induced pluripotent stem cells (hiPSCs) represent a prime candidate cell type for current research and future cell therapy because of their significant self-renewal, differentiation potential and the relative lack of ethical conflict. With the advent of efficient technology of reprogramming peripheral blood mononuclear cells (PBMCs) into hiPSCs, researchers can generate personalized lines of cells from which it will be possible to obtain differentiated cells in a less invasive way, introducing opportunities in treating diseases that are now considered incurable.

Until very recently, little success has been achieved in terms of skeletal muscle differentiation from hiPSCs. The purpose of this study is to explore the applicability of the differentiation into skeletal muscle progenitor cells from hiPSC cell lines and the associated biomolecular messages. It is anticipated that the derived skeletal muscle progenitor cells can be reprogrammed from PBMCs of female patients with urinary incontinence and/or pelvic organ prolapse and used in preclinical testing for relieving female urogenital problems.

ELIGIBILITY:
Inclusion Criteria:

* human induced pluripotent stem cells, hiPSCs

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cell lines (human induced pluripotent stem cells, hiPSCs)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Cell count | Day 50